CLINICAL TRIAL: NCT02763540
Title: Le rôle de la Cryobiopsie Transbronchique Dans le Diagnostic Des Maladies Pulmoniares Interstitielles
Brief Title: Pathological Comparisons of Surgical Open Lung Biopsies and Cryobiopsies in Non-IPF ILD
Acronym: CryoPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9607; 2015-A01350-49 (Other: RCB number)
Record Dates: First submitted 2016-04-13; First posted 2016-05-05 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Non Definite IPF; Interstitial Lung Diseases
Keywords: ILD; Pathology; diagnosis; lung biopsy
MeSH Terms: conditions — Lung Diseases, Interstitial; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lung cryobiopsy (Other)
  Interventions: Procedure: Lung cryobiopsy

INTERVENTIONS:
Procedure: Lung cryobiopsy — Transbronchial cryobiopsy
  Other Names: Per endoscopy

SUMMARY:
Pathological comparisons of surgical open lung biopsies and cryobiopsies in non-IPF ILD. Patients with non-IPF ILD eligible for an open lung biopsy will undergo cryobiopsy in the same time. Between observers agreement will be assessed for each pairs of samples.

ELIGIBILITY:
Inclusion Criteria:

* Non IPF ILD eligible for surgical lung biopsy reviewed during multidisciplinary approach

Exclusion Criteria:

* Ineligible for lung biopsy: pulmonary hypertension, coagulation deficiency, FEV<11, giant emphysematous bullae, hemodynamic instability severe hypoxia, general anesthetic ineligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
The percentage of concordant diagnoses between cryobiopsy and surgical lung biopsy. | for statistical analysis, 12 months after the first inclusion
  The gold standard is the consensual diagnosis between the two readers established from surgical biopsy

SECONDARY OUTCOMES:
The percentage homology between diagnosis obtained by surgical biopsy and cryobiopsy with the multidisciplinary approach | one day after inclusion
The percentage homology intra and inter observer for histopathological analysis of each type of sample by Mac Nemar test | for statistical analysis, 12 months after the first inclusion
The number of elementary lesions actually present in the two samples for the same patient | One day after inclusion
The time of the gesture and the respective anesthetic complexities of each procedure | One day after inclusion
The rate of adverse events | for statistical analysis, 12 months after the first inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bourdin, MD, PhD, Principal Investigator — University Hospitals of Montpellier
Locations (2):
- Arnaud de Villeneuve University Hospital, Montpellier, France
- S'Orsola-Malpighi hospital, Bologna, Italy

REFERENCES:
- [Background] Romagnoli M, Colby TV, Suehs CM, Vachier I, Molinari N, Bourdin A. Cryobiopsy Compared with Surgical Lung Biopsy in ILD: Reply to Maldonado et al., Froidure et al., Bendstrup et al., Agarwal et al., Richeldi et al., Rajchgot et al., and Quadrelli et al. Am J Respir Crit Care Med. 2019 Oct 1;200(7):944-946. doi: 10.1164/rccm.201906-1252LE. No abstract available. PMID 31442081
- [Background] Bourdin A, Suehs CM, Colby TV, Vachier I, Molinari N, Romagnoli M. Reply to Wand et al.: Role of Transbronchial Cryobiopsy in Interstitial Lung Diseases: An Ongoing Tale. Am J Respir Crit Care Med. 2020 Jan 15;201(2):260-261. doi: 10.1164/rccm.201909-1736LE. No abstract available. PMID 31535900
- [Background] Bourdin A, Romagnoli M, Gamez AS, Hireche K, Berthet JP, Mallet JP, Vachier I, Nava S, Reynaud P, Molinari N, Suehs C. Careful consideration of the bleeding caused by transbronchial lung cryobiopsies. Eur Respir J. 2020 May 21;55(5):1902415. doi: 10.1183/13993003.02415-2019. Print 2020 May. No abstract available. PMID 32439734
- [Result] Romagnoli M, Colby TV, Berthet JP, Gamez AS, Mallet JP, Serre I, Cancellieri A, Cavazza A, Solovei L, Dell'Amore A, Dolci G, Guerrieri A, Reynaud P, Bommart S, Zompatori M, Dalpiaz G, Nava S, Trisolini R, Suehs CM, Vachier I, Molinari N, Bourdin A. Poor Concordance between Sequential Transbronchial Lung Cryobiopsy and Surgical Lung Biopsy in the Diagnosis of Diffuse Interstitial Lung Diseases. Am J Respir Crit Care Med. 2019 May 15;199(10):1249-1256. doi: 10.1164/rccm.201810-1947OC. PMID 30864813
- [Result] Suehs C, Bourdin A, Vachier I, Molinari N, Romagnoli M. Transbronchial cryobiopsy in the diagnosis of interstitial lung diseases: methodologies and perspectives from the Cryo-PID and COLDICE studies. Ann Transl Med. 2020 Oct;8(20):1330. doi: 10.21037/atm-20-2814. No abstract available. PMID 33209910
- [Result] Reynaud P, Ahmed E, Serre I, Knabe L, Bommart S, Suehs C, Vachier I, Berthet JP, Romagnoli M, Vernisse C, Mallet JP, Gamez AS, Bourdin A. Club Cell Loss as a Feature of Bronchiolization in ILD. Front Immunol. 2021 Feb 26;12:630096. doi: 10.3389/fimmu.2021.630096. eCollection 2021. PMID 33717159